CLINICAL TRIAL: NCT01744314
Title: Indomethacin Prophylaxis for Heterotopic Ossification After Surgical Treatment of Elbow Trauma: A Randomized Prospective Double-blinded Study.
Brief Title: Indomethacin Prophylaxis for Heterotopic Ossification After Surgical Treatment of Elbow Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, George Athwal, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102903
Record Dates: First submitted 2012-11-19; First posted 2012-12-06 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Elbow Trauma Requiring Operative Management
Keywords: Elbow trauma,Heterotopic Ossification,Indomethacin, Prophylaxis
MeSH Terms: interventions — Indomethacin; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- drug (Experimental): The treatment arm will receive 21 days of Indomethacin and Pantoprazole (gastrointestinal protective agent). The patients will receive Indomethacin 25mg three times a day and Pantoprozole 40mg once a day.
  Interventions: Drug: Indomethacin and Pantoprazole
- placebo (Placebo Comparator): The placebo group will receive microcrystalline cellulose powder tablets to be taken as a control. The placebo will be dosed at the same intervals and duration as the treatment arm in this study.
  Interventions: Drug: microcrystalline cellulose powder tablets

INTERVENTIONS:
Drug: Indomethacin and Pantoprazole
  Arms: drug
Drug: microcrystalline cellulose powder tablets
  Arms: placebo

SUMMARY:
Patients who present to our institution with a traumatic injury to their elbow who need operative management will be randomized to one of two groups; a treatment arm and a control arm. The treatment arm will receive a three-week postoperative course of indomethacin while the control group will not. We will follow both groups to assess whether or not indomethacin prophylaxis affects the rate of heterotopic ossification.

ELIGIBILITY:
Inclusion Criteria:

* Terrible Triad
* Radial head fracture surgical treatment
* Monteggia and Trans-olecranon Fracture Dislocations
* Distal Biceps Tendon Injuries
* Distal Humerus Fractures
* Coronoid Fractures
* Capitellar-Trochlear fractures
* Olecranon Fractures

Exclusion Criteria:

* Associated Traumatic Brain Injury
* Burn Injuries associated with elbow trauma
* History of Gastric Ulcers
* Documented allergies to any Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)
* Severe Asthma
* Previous operative fixation to affected elbow
* Participation in other research study
* Inability to speak / understand English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
change in post operative radiographic evaluation | 6 weeks and 3, 6 and 12 mfup
  AS a standard care patients will be routinely assess at three, six , twelve and twenty four months post-operatively.

SECONDARY OUTCOMES:
change in range of motion | 6 weeks and 3, 6 and 12 mfup
  measuring range of motion with a goniometer will be performed at 6 weeks and 3, 6 and 12 mfup
Patient Rate Elbow Evaluation | 6 weeks and 3, 6 and 12 mfup
  is a 20-item questionnaire designed to measure elbow pain and disability
The Mayo Elbow Performance score | 6 weeks and 3, 6 and 12 mfup
  is an instrument used to test the limitations to use the elbow during ADL caused by the pathology
Disabilities of the Arm, Shoulder and Hand | 6 weeks and 3, 6 and 12 mfup
  is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb.

CONTACTS AND LOCATIONS:
Locations (1):
- HULC, St Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- See also: Canadian Orthopaedic Association — http://www.coa-aco.org/